CLINICAL TRIAL: NCT07106372
Title: A Multi-center, Single-arm, Open-label Study to Evaluate the Safety and Efficacy of Stapokibatrt in Children With Atopic Dermatitis
Brief Title: A Study of Stapokibatrt in Children Subjects With Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM310-101218
Record Dates: First submitted 2025-08-05; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stapokibatrt group (Experimental)
  Interventions: Biological: Stapokibatrt

INTERVENTIONS:
Biological: Stapokibatrt — Stapokibatrt Subcutaneous injection

SUMMARY:
This is a multi-center, single-arm, open-label phase 3 study to evaluate the safety, efficacy, Pharmacokinetics(PK) and immunogenicity of Stapokibatrt in children with Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the continuing study and sign the written Informed Consent Form(ICF).
* Subjects who must complete the evaluation of Week 18 of the main study.
* Have the ability to communicate well with the researcher and comply with the follow-up visits of the protocol.

Exclusion Criteria:

* Planned major surgical procedure during the patient's participation in this study.
* Any other circumstances in which the researcher deems not suitable to participate in this study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to week 44
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ma, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital Capital Medical University, Beijing, Beijing Municipality, China